CLINICAL TRIAL: NCT01085890
Title: Hypertension in Primary Health Care: Can More Intensive Work With Lifestyle Change Help Patients Achieve Blood Pressure Goals?
Brief Title: Hypertension in Primary Health Care: Lifestyle Change and Blood Pressure Goals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Lena Holm, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI 2006/1285-31; 511025-2672 (Other Grant/Funding Number: Stockholm County Council)
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Blood Pressure; Life Style
Keywords: Blood Pressure; Life Style; Body Mass Index; Obesity, Abdominal; Blood Chemical Analysis
MeSH Terms: conditions — Obesity, Abdominal | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing group (Experimental): The participants in this arm had 2 group seminars with information on hypertension and related lifestyle factors. They participated in 2 follow-up visits in which blood pressure was measured and motivational interviewing took place. The motivational interviewing focused on lifestyle factors, including physical activity, stress, tobacco use, alcohol habits, and diet.
  Interventions: Behavioral: Motivational interviewing
- Treatment as usual (No Intervention): Participants in this group received treatment as usual for their high blood pressure, but no informational seminars and no extra visits with motivational interviewing and blood pressure measurement.

INTERVENTIONS:
Behavioral: Motivational interviewing — The intervention consisted of 2 group seminars with information on hypertension and related lifestyle factors and 2 follow-up visits in which blood pressure was measured and motivational interviewing took place. The motivational interviewing focused on lifestyle factors, including physical activity, stress, tobacco use, alcohol habits, and diet.
  Arms: Motivational interviewing group

SUMMARY:
The purpose of this study is to determine whether a program that includes 1) group seminars and 2) follow-up visits with blood pressure measurement and motivational interviewing (MI) that is focused on lifestyle change affect blood pressure.

DETAILED DESCRIPTION:
High blood pressure is common in the population. In an earlier study conducted in our local geographical area, "How is health in Jordbro?" 46% of participants had a systolic blood pressure of >140 millimeters of mercury (mm Hg) and 22% had a diastolic blood pressure >90 mm Hg. 84% of those with known hypertension had a systolic blood pressure of >140. We thus found that many people in our area have heightened blood pressure, and hypothesized that many of these people, particularly those with mild hypertension, probably could be helped with lifestyle-related intervention.

All persons who came to Jordbro Primary Health Care Center during a 6-month period were invited to participate in the current study, and local press announcements were used to recruit additional participants. A total of 301 persons volunteered to participate. A total of 141 of the volunteers had a systolic blood pressure =>140 and/or a diastolic blood pressure of =>90, and these people became the study population. The 141 persons in the study population filled in a questionnaire with general background and lifestyle questions.

Of the 141 persons in the study population, 75 had previously known hypertension and 66 had hypertension that was previously unknown. Participants were then randomized such that an equal number of persons with previously known and previously unknown hypertension were included in a) a treatment group and b) a control group. Background information such as height, weight, pulse, smoking habits, other diseases, and prescription drugs was gathered. Blood sugar and lipid tests were conducted. Participants' family physician were contacted as necessary (e.g., if blood pressure was dangerously high).

The intervention consisted of 2 group seminars with information on hypertension and related lifestyle factors and 2 follow-up visits with each participant in which blood pressure was measured and motivational interviewing took place. The motivational interviewing focused on lifestyle factors, including physical activity, stress, tobacco use, alcohol habits, and diet. After 6 months, a follow-up was done that included blood pressure measurement and completion of the same questionnaire that was filled in at baseline.

ELIGIBILITY:
Inclusion Criteria:

* => 30 years
* ability to speak Swedish well enough to fill the baseline and follow-up questionnaires, participate in the seminars, and participate in the motivational interviewing

Exclusion Criteria:

* < 30 years
* inability to speak Swedish well enough to fill the baseline and follow-up questionnaires, participate in the seminars, and participate in the motivational interviewing

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 6 months after conclusion of study

SECONDARY OUTCOMES:
Lifestyle factors | 6 months after conclusion of study
  Lifestyle factors included physical activity, stress, tobacco use, alohol habits, and diet.
Body mass index (BMI) | 6 months after conclusion of study
  Body mass index = weight in kilograms/height in square meters
Abdominal circumference | 6 months after conclusion of study
  Measurement in centimeters of the abdomen.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Holm, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Jordbro Primary Health Care Center, Haninge, Sweden

REFERENCES:
- [Background] Al-Windi A. Detection and treatment of hypertension in general health-care practice: a patient-based study. J Hum Hypertens. 2005 Oct;19(10):775-86. doi: 10.1038/sj.jhh.1001902. PMID 15988540
- [Background] Al-Windi A. The validity of a questionnaire on medicines used in health care practice: comparison of a questionnaire and computerized medical record survey. Eur J Clin Pharmacol. 2003 Aug;59(4):321-9. doi: 10.1007/s00228-003-0615-1. Epub 2003 Jul 4. PMID 12845507